CLINICAL TRIAL: NCT01082068
Title: A Phase 1/2 Dose-Escalation Study of XL147 (SAR245408) or XL765 (SAR245409) in Combination With Letrozole in Subjects With Hormone Receptor-Positive and HER2-Negative Breast Cancer Refractory to a Nonsteroidal Aromatase Inhibitor
Brief Title: Study of XL147 (SAR245408) or XL765 (SAR245409) in Combination With Letrozole in Subjects With Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARD11437; XL147-202 (Other: (Other study code))
Record Dates: First submitted 2010-03-04; First posted 2010-03-08 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: HER2 negative; Hormone Receptor Positive; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — XL147; XL765; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): XL147 (SAR245408) + letrozole
  Interventions: Drug: XL147 (SAR245408); Drug: letrozole (Femara)
- Arm 2 (Experimental): XL765 + letrozole
  Interventions: Drug: XL765 (SAR245409); Drug: letrozole (Femara)

INTERVENTIONS:
Drug: XL147 (SAR245408) — given orally once daily as tablets
  Arms: Arm 1
Drug: XL765 (SAR245409) — given orally twice daily as capsules
  Arms: Arm 2
Drug: letrozole (Femara) — given orally once daily as tablets

SUMMARY:
Phase 1 of this study will evaluate the maximum tolerated dose (MTD) of XL147 when given in combination with letrozole (Femara) and of XL765 when given in combination with letrozole. After the MTD is established for each combination (Phase 2), subjects will be enrolled to evaluate the preliminary efficacy and safety of these combinations in subjects with breast cancer refractory to a non-steroidal aromatase inhibitor that is ER+/PGR+ and HER2-. Letrozole is used in the treatment of different types of breast cancer, but patients can develop resistance.

Upregulation of PI3K activity is one of the most common characteristics of human cancer cells, including breast tumor cells. Activation of PI3K results in stimulation of AKT and mTOR kinases, resulting in the promotion of tumor cell proliferation and survival. Preclinical and retrospective clinical data suggest that aberrant activation of the PI3K pathway may play a role in aromatase inhibitor resistance in patients with ER+, HER2- breast cancer. XL147 is a potent inhibitor of PI3K, and XL765 is a potent dual inhibitor of PI3K and mTOR; therefore either of these compounds in combination with letrozole warrants clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* The subject has histologically confirmed breast cancer that is ER+ and/or PGR+.
* The subject's breast cancer is negative for HER2.
* The subject has recurrent or metastatic breast cancer that is refractory to a nonsteroidal aromatase inhibitor and has either disease progression or disease recurrence.
* Subjects previously treated with letrozole must be able to tolerate the approved dose and schedule of letrozole.
* For subjects enrolled in Phase 2, either archival tumor samples must be available, or the subject must be willing to undergo a fresh biopsy.
* In Phase 2, at least 30 subjects in each arm must have measurable disease
* The subject is a postmenopausal female.
* If a subject is currently receiving bisphosphonates, the subject must have received the bisphosphonates for at least 2 months before starting study treatment.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
* The subject has adequate organ and marrow function.
* The subject has no other diagnosis of malignancy or evidence of other malignancy for 2 years before screening for this study (except non-melanoma skin cancer or in situ carcinoma of the cervix).
* The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document.

Exclusion Criteria:

* The subject has received prior treatment with a selective inhibitor of PI3K, AKT, and/or mTOR.
* Certain restrictions on prior therapies apply.
* The subject has not recovered from toxicity due to prior therapy to Grade ≤ 1 or to pre-therapy baseline.
* The subject has untreated, symptomatic, or progressive brain metastases.
* The subject has only non-measurable lesions, other than bone, skin, or chest wall metastasis
* The subject has to start cytotoxic chemotherapy due to rapid progressive disease involving major organs.
* The subject has prothrombin time/ International Normalized Ratio (PT/ INR) or partial thromboplastin time (PTT) test results at screening that are above 1.3 x the laboratory upper limit of normal.
* The subject has uncontrolled significant intercurrent illness.
* The subject has a baseline corrected QT interval (QTc) > 470 ms.
* The subject has a diagnosis of uncontrolled diabetes mellitus.
* The subject is known to be positive for the human immunodeficiency virus (HIV).
* The subject has a previously identified allergy or hypersensitivity to components of the study treatment formulation(s).
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of XL147 and letrozole and XL765 and letrozole | at weekly and bi-weekly study visits
In Phase 1, to determine the maximum tolerated dose of XL147 in combination with letrozole and of XL765 in combination with letrozole | assessed by weekly study visits
In Phase 2, to evaluate progression-free survival at 3 months | tumor assessments at Week 13 and every 8 weeks thereafter

SECONDARY OUTCOMES:
In Phase 2, to assess other clinical benefit and efficacy parameters | tumor assessments at Week 13 and every 8 weeks thereafter
Pharmacokinetics and pharmacodynamics of XL147, XL765 and letrozole | assessed every 2 weeks, then every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (17):
- United States (11):
  - Investigational Site Number 1537, Los Angeles, California
  - Investigational Site Number 1601, Denver, Colorado
  - Investigational Site Number 1238, Fort Meyers, Florida
  - Investigational Site Number 1441, Chicago, Illinois
  - Investigational Site Number 1138, Boston, Massachusetts
  - Investigational Site Number 1331, Ann Arbor, Michigan
  - Investigational Site Number 1330, Detroit, Michigan
  - Investigational Site Number 5201, Columbia, Missouri
  - Investigational Site Number 1252, Durham, North Carolina
  - Investigational Site Number 1214, Nashville, Tennessee
  - Investigational Site Number 5246, El Paso, Texas
- France (2):
  - Investigational Site Number 3321, Nantes Saint Herblain
  - Investigational Site Number 3324, Paris
- Spain (4):
  - Investigational Site Number 3415, Barcelona
  - Investigational Site Number 3419, Barcelona
  - Investigational Site Number 3413, Madrid
  - Investigational Site Number 3420, Madrid